CLINICAL TRIAL: NCT00976339
Title: Pilot Biomarker Modulation Study of Vitamin D in Premenopausal Women at High Risk for Breast Cancer
Brief Title: Study of Vitamin D for Premenopausal Women at High Risk for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Katherine D. Crew (Other)
Collaborators: Prevent Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Katherine D. Crew, Florence Irving Assistant Professor of Medicine and Assistant Professor of Epidemiology, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAC3089
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Vitamin D; Premenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cholecalciferol 20,000 IU (Experimental): Participants will receive Cholecalciferol 20,000 IU (2 capsules) weekly for one year.
  Interventions: Drug: Cholecalciferol
- Cholecalciferol 30,000 IU (Experimental): Participants will receive Cholecalciferol 30,000 IU (3 capsules) weekly for one year.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol is a vitamin D3. Vitamin D is important for the absorption of calcium from the stomach and for the functioning of calcium in the body. Cholecalciferol is used to treat or prevent many conditions caused by a lack of vitamin D.
  Cholecalciferol will be available in gel capsule form at 10,000 IU (0.25 mg cholecalciferol) each.
  Other Names: Vitamin D3

SUMMARY:
This proposal is for a pilot study of 20 premenopausal women at high risk for breast cancer development who will receive high dose vitamin D3, cholecalciferol 20,000 IU (2 capsules) weekly, or 30,000 IU (3 capsules) weekly, for 1 year. The primary objective of this study is to determine the feasibility of a 1-year intervention of vitamin D in this study population. Secondary objectives include evaluating the biologic effects of vitamin D supplementation on blood based and image-based biomarkers.

DETAILED DESCRIPTION:
Vitamin D has diverse biological effects relevant to carcinogenesis, including known cross-talk between the vitamin D receptor (VDR) and insulin-like growth factor (IGF) signaling pathways. Based upon observational data, women with serum 25(OH) D levels greater than 40-50 ng/ml had a 50% lower risk of breast cancer compared to women with vitamin D deficiency.

Vitamin D is a fat-soluble vitamin which is produced in the body and may come from food sources. Epidemiologic studies suggest that vitamin D may influence breast cancer development, which has resulted in increased interest in the use of vitamin D for the treatment and prevention of breast cancer. Numerous experimental studies have shown that vitamin D compounds have anti-carcinogenic properties against breast cancer. Given the epidemiologic data and the extensive preclinical evidence of the anti-tumor effects of vitamin D, it is therefore reasonable to test the biological effects of high-dose vitamin D in early phase clinical trials. The investigators hypothesize that vitamin D3, cholecalciferol, will modulate biomarkers of breast cancer risk.

The relationship between vitamin D status and mammographic density (MD), a strong predictor of breast cancer risk, remains unclear [8]. MD refers to the relative proportions of radiolucent fat and radiodense epithelial and stromal tissue and may serve as a useful intermediate biomarker for breast cancer risk assessment in investigations of potential chemopreventive agents. Cross-sectional studies evaluating the association between vitamin D intake and MD observed an inverse association among premenopausal women, particularly with high serum IGF-1 and low serum IGF binding protein-3 (IGFBP-3). However, there is limited data on the biologic effects of vitamin D supplementation for breast cancer prevention in human intervention trials.

ELIGIBILITY:
Inclusion Criteria:

* Elevated risk of breast cancer defined as having at least one of the following: (1) Predicted 5-year modified Gail model risk of 1.7% or greater, (2) Lobular carcinoma in situ, (3) Known BRCA1 or BRCA2 deleterious mutation carrier, (4) Prior history of ductal carcinoma in situ, if no current tamoxifen use or prior radiation to the contralateral breast.
* Age 21 years or older.
* Premenopausal defined as < 6 months since the last menstrual period, no prior bilateral oophorectomy, not on estrogen replacement, and serum Follicle-stimulating hormone (FSH) values consistent with institutional normal values for the premenopausal state.
* Normal breast exam and mammogram (BIRADS score of 1 or 2).
* Baseline mammographic density ≥25% as assessed qualitatively by the mammographer (25-50% = "scattered fibroglandular densities"; >50-75% = "heterogeneously dense breasts"; >75% = "extremely dense breasts").
* Baseline serum 25-hydroxyvitamin D <32 ng/ml.
* Prior tamoxifen use is allowed provided treatment is discontinued at least 28 days prior to enrollment.
* Willingness to allow submission of core needle breast biopsy for pathology review and collection of blood for biomarker analysis and banking.
* At least one breast available for imaging and biopsy.
* Willingness to not take calcium or vitamin D supplements during the one year intervention, due to the potential risk of hypercalcemia/hypercalciuria with high dose vitamin D. Premenopausal women who need to take calcium supplementation for any medical condition will be excluded from the study. Dietary restrictions on calcium intake may be imposed if the subject is found to have borderline high serum or urine levels of calcium during the study intervention and a list of dietary sources of calcium will be provided.
* Normal serum calcium.
* No history of kidney stones.
* Adequate renal and hepatic function: serum creatinine, bilirubin, aspartate aminotransferase (AST), alanine transaminase (ALT) and alkaline phosphatase < 2.0 x the institutional upper limit of normal (IULN).
* No hypersensitivity reactions to vitamin D.
* Performance status of 0 or 1.
* Not pregnant or nursing.
* Agree to use effective contraception, hormone-based oral contraceptives allowed but switching birth control methods is discouraged while on-study.
* No significant medical or psychiatric condition that would preclude study completion.

Exclusion Criteria:

* Not meeting one or any of inclusion criteria

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Crew, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center Herbert Irving Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vieth R. Critique of the considerations for establishing the tolerable upper intake level for vitamin D: critical need for revision upwards. J Nutr. 2006 Apr;136(4):1117-22. doi: 10.1093/jn/136.4.1117. PMID 16549491
- [Background] Vieth R, Chan PC, MacFarlane GD. Efficacy and safety of vitamin D3 intake exceeding the lowest observed adverse effect level. Am J Clin Nutr. 2001 Feb;73(2):288-94. doi: 10.1093/ajcn/73.2.288. PMID 11157326
- [Background] Vieth R. Vitamin D supplementation, 25-hydroxyvitamin D concentrations, and safety. Am J Clin Nutr. 1999 May;69(5):842-56. doi: 10.1093/ajcn/69.5.842. PMID 10232622
- [Background] Garland CF, Garland FC, Gorham ED, Lipkin M, Newmark H, Mohr SB, Holick MF. The role of vitamin D in cancer prevention. Am J Public Health. 2006 Feb;96(2):252-61. doi: 10.2105/AJPH.2004.045260. Epub 2005 Dec 27. PMID 16380576
- [Background] Bertone-Johnson ER, Chen WY, Holick MF, Hollis BW, Colditz GA, Willett WC, Hankinson SE. Plasma 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D and risk of breast cancer. Cancer Epidemiol Biomarkers Prev. 2005 Aug;14(8):1991-7. doi: 10.1158/1055-9965.EPI-04-0722. PMID 16103450
- [Background] John EM, Schwartz GG, Dreon DM, Koo J. Vitamin D and breast cancer risk: the NHANES I Epidemiologic follow-up study, 1971-1975 to 1992. National Health and Nutrition Examination Survey. Cancer Epidemiol Biomarkers Prev. 1999 May;8(5):399-406. PMID 10350434
- [Background] Shin MH, Holmes MD, Hankinson SE, Wu K, Colditz GA, Willett WC. Intake of dairy products, calcium, and vitamin d and risk of breast cancer. J Natl Cancer Inst. 2002 Sep 4;94(17):1301-11. doi: 10.1093/jnci/94.17.1301. PMID 12208895
- [Background] Lowe LC, Guy M, Mansi JL, Peckitt C, Bliss J, Wilson RG, Colston KW. Plasma 25-hydroxy vitamin D concentrations, vitamin D receptor genotype and breast cancer risk in a UK Caucasian population. Eur J Cancer. 2005 May;41(8):1164-9. doi: 10.1016/j.ejca.2005.01.017. Epub 2005 Apr 14. PMID 15911240
- [Background] Chen WY, Bertone-Johnson ER, Hunter DJ, Willett WC, Hankinson SE. Associations between polymorphisms in the vitamin D receptor and breast cancer risk. Cancer Epidemiol Biomarkers Prev. 2005 Oct;14(10):2335-9. doi: 10.1158/1055-9965.EPI-05-0283. PMID 16214913
- [Background] Narvaez CJ, Zinser G, Welsh J. Functions of 1alpha,25-dihydroxyvitamin D(3) in mammary gland: from normal development to breast cancer. Steroids. 2001 Mar-May;66(3-5):301-8. doi: 10.1016/s0039-128x(00)00202-6. PMID 11179738
- [Background] Mathiasen IS, Sergeev IN, Bastholm L, Elling F, Norman AW, Jaattela M. Calcium and calpain as key mediators of apoptosis-like death induced by vitamin D compounds in breast cancer cells. J Biol Chem. 2002 Aug 23;277(34):30738-45. doi: 10.1074/jbc.M201558200. Epub 2002 Jun 18. PMID 12072431
- [Background] Brenner BM, Russell N, Albrecht S, Davies RJ. The effect of dietary vitamin D3 on the intracellular calcium gradient in mammalian colonic crypts. Cancer Lett. 1998 May 15;127(1-2):43-53. doi: 10.1016/s0304-3835(98)00005-6. PMID 9619857
- [Background] Lowe L, Hansen CM, Senaratne S, Colston KW. Mechanisms implicated in the growth regulatory effects of vitamin D compounds in breast cancer cells. Recent Results Cancer Res. 2003;164:99-110. doi: 10.1007/978-3-642-55580-0_6. PMID 12908448
- [Background] Welsh J. Vitamin D and breast cancer: insights from animal models. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1721S-4S. doi: 10.1093/ajcn/80.6.1721S. PMID 15585794
- [Background] Wolfe JN. Breast patterns as an index of risk for developing breast cancer. AJR Am J Roentgenol. 1976 Jun;126(6):1130-7. doi: 10.2214/ajr.126.6.1130. PMID 179369
- [Background] Boyd NF, Lockwood GA, Byng JW, Tritchler DL, Yaffe MJ. Mammographic densities and breast cancer risk. Cancer Epidemiol Biomarkers Prev. 1998 Dec;7(12):1133-44. PMID 9865433
- [Background] Lee NA, Rusinek H, Weinreb J, Chandra R, Toth H, Singer C, Newstead G. Fatty and fibroglandular tissue volumes in the breasts of women 20-83 years old: comparison of X-ray mammography and computer-assisted MR imaging. AJR Am J Roentgenol. 1997 Feb;168(2):501-6. doi: 10.2214/ajr.168.2.9016235.
- [Background] Heywang-Kobrunner SH, Viehweg P, Heinig A, Kuchler C. Contrast-enhanced MRI of the breast: accuracy, value, controversies, solutions. Eur J Radiol. 1997 Feb;24(2):94-108. doi: 10.1016/s0720-048x(96)01142-4. PMID 9097051
- [Background] Eng-Wong J, Orzano-Birgani J, Chow CK, Venzon D, Yao J, Galbo CE, Zujewski JA, Prindiville S. Effect of raloxifene on mammographic density and breast magnetic resonance imaging in premenopausal women at increased risk for breast cancer. Cancer Epidemiol Biomarkers Prev. 2008 Jul;17(7):1696-701. doi: 10.1158/1055-9965.EPI-07-2752. Epub 2008 Jun 26. PMID 18583470
- [Background] Arai M, Sasaki A, Saito N, Nakazato Y. Immunohistochemical analysis of cleaved caspase-3 detects high level of apoptosis frequently in diffuse large B-cell lymphomas of the central nervous system. Pathol Int. 2005 Mar;55(3):122-9. doi: 10.1111/j.1440-1827.2005.01808.x. PMID 15743320
- [Background] Lensmeyer GL, Wiebe DA, Binkley N, Drezner MK. HPLC method for 25-hydroxyvitamin D measurement: comparison with contemporary assays. Clin Chem. 2006 Jun;52(6):1120-6. doi: 10.1373/clinchem.2005.064956. Epub 2006 Mar 30. PMID 16574756
- [Background] Gao P, Scheibel S, D'Amour P, John MR, Rao SD, Schmidt-Gayk H, Cantor TL. Development of a novel immunoradiometric assay exclusively for biologically active whole parathyroid hormone 1-84: implications for improvement of accurate assessment of parathyroid function. J Bone Miner Res. 2001 Apr;16(4):605-14. doi: 10.1359/jbmr.2001.16.4.605. PMID 11315988
- [Background] Lee LG, Connell CR, Bloch W. Allelic discrimination by nick-translation PCR with fluorogenic probes. Nucleic Acids Res. 1993 Aug 11;21(16):3761-6. doi: 10.1093/nar/21.16.3761. PMID 8367293
- [Background] Hershman, D. L., McMahon, D., Irani, D., Cucchiara, G., Crew, K. D., Raptis, G., and Shane, E. High prevalence of vitamin D deficiency in premenopausal women with early-stage breast cancer. Proc Am Soc Clin Oncol, pp. Abst #8568. Atlanta, 2006.
- [Background] Chlebowski, R. T., Johnson, K. C., Kooperberg, C., Hubbell, A., Lane, D., O'Sullivan, M., Cummings, S., Rohan, T., Khandekar, J., and Investigators, T. W. s. H. I. The Women's Health Initiative randomized trial of calcium plus vitamin D: effects on breast cancer and arthralgias. Proceedings of the American Society of Clinical Oncology 24, pp. LBA6. Atlanta, 2006.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Referrals to the Columbia breast oncology clinic for breast cancer chemoprevention will be recruited medical oncologist or via recruitment flyers. Recruitment letters will be sent to high-risk women who participated in the Metropolitan Breast Cancer Family Registry and Women at Risk (WAR) database.
Groups:
- Cholecalciferol 20,000 IU: Subjects received Cholecalciferol 20,000 IU weekly for 1 year.
- Cholecalciferol 30,000 IU: Subjects received Cholecalciferol 30,000 IU weekly for one year
Period: Overall Study
Arm/Group | Cholecalciferol 20,000 IU | Cholecalciferol 30,000 IU
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cholecalciferol 20,000 IU: Subjects received Cholecalciferol 20,000 IU weekly, for 1 year
- Cholecalciferol 30,000 IU: Subjects received Cholecalciferol 30,000 IU weekly, for 1 year
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol 20,000 IU | Cholecalciferol 30,000 IU | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Count of Participants; unit: Participants]
  > 21 years | 10 | 10 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Successfully Completed the 1-year Intervention
Time Frame: 1 year
Population: Data for this study (NCT00976339) is combined with the data for another study (NCT00859651); see NCT00859651 for combined results. Investigator is unable to determine the subject data that should be entered for this study alone, since subject data was combined for the purpose of data analysis. Data for this study alone was not analyzed.
Groups:
- Cholecalciferol 20,000 IU: Subjects received Cholecalciferol 20,000 IU weekly 1 year
- Cholecalciferol 30,000 IU: Subjects received Cholecalciferol 30,000 IU weekly 1 year
Arm/Group | Cholecalciferol 20,000 IU | Cholecalciferol 30,000 IU
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Mammographic Breast Density
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Cholecalciferol 20,000 IU | Cholecalciferol 30,000 IU
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Data for this study (NCT00976339) is combined with the data for another study (NCT00859651); see NCT00859651 for combined results. Investigator is unable to determine the subject data that should be entered for this study alone, since subject data was combined for the purpose of data analysis. Data for this study alone was not analyzed.
Arm/Group | Cholecalciferol 20,000 IU | Cholecalciferol 30,000 IU
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Data for this study (NCT00976339) is combined with the data for another study (NCT00859651); see NCT00859651 for combined results. Data for this study alone was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No